CLINICAL TRIAL: NCT02929069
Title: A Unified Intervention for Young Gay and Bisexual Men's Minority Stress, Mental Health, and HIV Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1509016430; 1R01MH109413-01 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome
Keywords: Minority Stress
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ESTEEM (Experimental): Participants in all arms will receive Voluntary Counselling and Testing (VCT). Participants randomized to this arm will receive ESTEEM. ESTEEM is a 10-session intervention based on the Unified Protocol,an individually-delivered CBT intervention with efficacy for reducing stress-sensitive mental health disorders (e.g., depression, anxiety) by enhancing emotion regulation skills; reducing avoidance patterns; and improving motivation and self-efficacy for behavior change.
  Interventions: Behavioral: ESTEEM; Behavioral: VCT
- Community Mental Health Treatment (CMHT) (Active Comparator): Participants in all arms will receive Voluntary Counselling and Testing (VCT). Participants randomized to this arm will receive Community Mental Health Treatment (CMHT). CMHT is the current standard of care for LGB individuals who seek mental, behavioral, or sexual health care is LGB-affirmative therapy.The practice of LGB-affirmative therapy is outlined across 21 guidelines published by the American Psychological Association.
  Interventions: Behavioral: CMHT; Behavioral: VCT
- Voluntary Counselling and Testing (VCT) (Active Comparator): Participants randomized to the VCT only arm will not receive any further intervention. VCT will be based on on CDC guidelines and the control arms of large community-based RCTs (e.g., Projects RESPECT, EXPLORE, AWARE). VCT will consist of one 45-minute session given that 1-session VCT is as effective as 2-session VCT for GBM.
  Interventions: Behavioral: VCT

INTERVENTIONS:
Behavioral: ESTEEM — ESTEEM is a 10-session intervention based on the Unified Protocol, an individually-delivered CBT intervention with efficacy for reducing stress-sensitive mental health disorders (e.g., depression, anxiety) by enhancing emotion regulation skills; reducing avoidance patterns; and improving motivation and self-efficacy for behavior change.
  Arms: ESTEEM
Behavioral: CMHT — CMHT is the current standard of care for LGB individuals who seek mental, behavioral, or sexual health care is LGB-affirmative therapy.The practice of LGB-affirmative therapy is outlined across 21 guidelines published by the American Psychological Association.
  Arms: Community Mental Health Treatment (CMHT)
Behavioral: VCT — Voluntary Counselling and Testing (VCT).

SUMMARY:
The intent of the proposed randomized controlled trial is to test the efficacy of a principle-based, transdiagnostic cognitive behavioral therapy (CBT) intervention that addresses the pathways through which minority stress compromises young gay and bisexual men's (YGBM) co-occurring mental (e.g., depression), behavioral (e.g., substance use), and sexual (e.g., condomless anal sex) health problems.

DETAILED DESCRIPTION:
ESTEEM (Effective Skills to Empower Effective Men) is a 10-session skills-building intervention designed to reduce young gay and bisexual men's (YGBM) co-occurring health risks by reducing the underlying cognitive, affective, and behavioral pathways through which minority stress impairs YGBM's health. ESTEEM is based on the Unified Protocol, a cognitive-behavioral therapy (CBT) approach with efficacy across mental health and risk behaviors. In an initial study to create ESTEEM , the Unified Protocol was adapted by conducting interviews with 21 YGBM-expert mental health providers and 20 depressed, anxious YGBM at high risk for HIV infection. In a preliminary trial (NCT02448186), ESTEEM significantly reduced YGBM's spectrum of interrelated health threats, making it the first evidence-based intervention to simultaneously improve mental health, substance use, and sexual health outcomes among YGBM.

Important questions remain in order to validate the efficacy and potential cost-effectiveness of ESTEEM. Accordingly, we propose a 3-arm RCT that would examine (1) whether ESTEEM (arm 1) demonstrates significant improvements compared to existing LGBT-affirmative community mental health treatment (CMHT; arm 2) or standard HIV/STD voluntary counseling and testing (VCT; arm 3) for high-risk depressed and anxious YGBM and (2) whether it improves outcomes through reducing hypothesized cognitive, affective, and behavioral minority stress processes.

ELIGIBILITY:
Inclusion Criteria:

* self-identification as a gay, bisexual or queer man;
* HIV-negative status confirmed through in-office testing;
* diagnosis of any DSM-5 depressive, anxiety, or trauma-/stress-related disorder;
* risk of HIV transmission through sexual activity (≥ 1 act of past-90-day-condomless anal sex involving a flesh penis with a partner with an unknown HIV status or an HIV-positive status, unless with an HIV-positive primary or main partner with known undetectable viral load or an HIV-negative primary or main partner who is known to be adherent to PrEP);
* not themselves currently adherent to PrEP (defined as taking PrEP on ≥ 4 days/week);
* NYC or Miami residential stability and planned availability for 12 months;
* English-language proficiency; and (9) provision of informed consent.

Exclusion Criteria:

* current active suicidality or homicidality (but not passive suicidality);
* evidence of active untreated mania, psychosis, or gross cognitive impairment;
* current enrollment in another intervention study;
* currently receiving 1 or more mental health treatment sessions/month or 8 or more CBT sessions within the past year;
* HIV-positive status (confirmed through in-office testing).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2016-09; Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, PhD, Principal Investigator — MYSM School Of Medicine
Locations (2):
- United States (2):
  - School of Public Health, Yale University, New Haven, Connecticut
  - Clinical Research Building, University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Keefe JR, Rodriguez-Seijas C, Jackson SD, Branstrom R, Harkness A, Safren SA, Hatzenbuehler ML, Pachankis JE. Moderators of LGBQ-affirmative cognitive behavioral therapy: ESTEEM is especially effective among Black and Latino sexual minority men. J Consult Clin Psychol. 2023 Mar;91(3):150-164. doi: 10.1037/ccp0000799. Epub 2023 Feb 13. PMID 36780265
- [Derived] Pachankis JE, McConocha EM, Reynolds JS, Winston R, Adeyinka O, Harkness A, Burton CL, Behari K, Sullivan TJ, Eldahan AI, Esserman DA, Hatzenbuehler ML, Safren SA. Project ESTEEM protocol: a randomized controlled trial of an LGBTQ-affirmative treatment for young adult sexual minority men's mental and sexual health. BMC Public Health. 2019 Aug 9;19(1):1086. doi: 10.1186/s12889-019-7346-4. PMID 31399071

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ESTEEM | Community Mental Health Treatment (CMHT) | Voluntary Counselling and Testing (VCT)
Started | 100 | 102 | 52
Completed 4 Month Follow Up | 83 | 76 | 43
Completed 8 Month Follow Up | 82 | 77 | 36
Assessed STI 12 Month | 74 | 75 | 38
Assessed HIV 12 Month | 76 | 76 | 39
Complete 12 Month Follow Up | 81 | 81 | 42
Completed | 81 | 81 | 42
Not Completed | 19 | 21 | 10

BASELINE CHARACTERISTICS:
Population: The total number of participants randomized was 254, but 1 participant dropped out following randomization and did not complete the baseline interview.
Groups:
- Community Mental Health Treatment (CMHT): Participants in all arms will receive Voluntary Counselling and Testing (VCT). Participants randomized to this arm will receive Community Mental Health Treatment (CMHT). CMHT is the current standard of care for LGB individuals who seek mental, behavioral, or sexual health care is LGB-affirmative therapy. The practice of LGB-affirmative therapy is outlined across 21 guidelines published by the American Psychological Association.
  One participant in this arm did not complete baseline measures and is thus excluded in the baseline measures section.
  CMHT: CMHT is the current standard of care for LGB individuals who seek mental, behavioral, or sexual health care is LGB-affirmative therapy.The practice of LGB-affirmative therapy is outlined across 21 guidelines published by the American Psychological Association.
  VCT: Voluntary Counselling and Testing (VCT).
- Total: Total of all reporting groups
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT) | Total
Number analyzed (Participants) | 100 | 52 | 101 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.31 (4.47) | 26.88 (3.43) | 26.6 (4.23) | 26.55 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 2 | 0 | 1 | 3
    Male | 98 | 52 | 100 | 250
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 24 | 41 | 108
  Not Hispanic or Latino | 57 | 28 | 60 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian /Alaskan Native | 1 | 0 | 0 | 1
  Asian | 5 | 2 | 3 | 10
  Black/African American | 20 | 2 | 21 | 43
  Multiracial | 12 | 12 | 14 | 38
  Native Hawaiian/Pacific Islander | 0 | 1 | 1 | 2
  White | 53 | 32 | 56 | 141
  Other | 9 | 3 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 100 | 52 | 101 | 253
Gender Identity [Count of Participants; unit: Participants] — Gender identity variable was "check all that apply;" percent out of total sample size denoted for each identity.
  Participants
    Man | 100 | 51 | 99 | 250
    Woman | 2 | 0 | 0 | 2
    Transgender Man | 2 | 0 | 0 | 2
    Genderqueer | 2 | 2 | 2 | 6
    Gender non-conforming/-binary | 2 | 0 | 1 | 3
    Two-spirit | 3 | 0 | 0 | 3
    Other | 1 | 0 | 1 | 2
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 25 | 9 | 19 | 53
  Gay | 69 | 39 | 78 | 186
  Queer | 6 | 4 | 3 | 13
  Uncertain | 0 | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  Less than College | 6 | 6 | 10 | 22
  College Degree | 94 | 46 | 91 | 231
Diagnoses [Count of Participants; unit: Participants] — All diagnoses presented, minus Substance-use disorder, were obtained using clinician-administered modules for listed disorders using the Mini-International Neuropsychiatric Interview for DSM-5 and ICD-10. Substance-use disorder was assessed for any of the following substance categories: stimulants, cocaine, opiates, hallucinogens, dissociatives, inhalants, cannabis, tranquilizers and miscellaneous.
  Participants
    Depression | 79 | 37 | 79 | 195
    Dysthymia | 33 | 9 | 40 | 82
    Panic Disorder | 16 | 12 | 25 | 53
    Agoraphobia | 24 | 11 | 25 | 60
    Social Anxiety Disorder | 37 | 20 | 49 | 106
    Obsessive Compulsive Disorder | 23 | 7 | 20 | 50
    Post-Traumatic Stress Disorder | 18 | 5 | 14 | 37
    Generalized Anxiety Disorder | 53 | 20 | 51 | 124
    Alcohol-Use Disorder | 27 | 13 | 22 | 62
    Substance-Use Disorder | 55 | 28 | 53 | 136

OUTCOME MEASURES:

1. Primary Outcome: Any Condomless Anal Sex Acts
Description: Our primary outcome is the presence (yes/no) of any condomless anal sex (CAS) in the absence of either PrEP or known undetectable viral load of HIV+ primary partners.The Time-Line Follow-Back Interview (TLFB) will be used to assess frequency of HIV risk behavior, including CAS, sex while under the influence of drugs or alcohol, and number of sexual partners, during the previous 3 months.
Time Frame: 8 Months
Population: Intention to Treat. One participant in each condition did not provide data for this outcome measure; overall number of participants analyzed does not include these participants.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Community Mental Health Treatment (CMHT) | Voluntary Counselling and Testing (VCT)
Number analyzed (Participants) | 81 | 76 | 35
Participants
  CAS = Yes | 43 | 47 | 17
  CAS = No | 38 | 29 | 18
Statistical Analysis 1: Comparison: ESTEEM vs Voluntary Counselling and Testing (VCT); Test type: Superiority; p = 0.52, Regression, Logistic; Risk Ratio (RR) = .88, 95% CI 2-sided [.52 to 1.25]

2. Secondary Outcome: Minority Stress: GRRS
Description: Assessments at baseline will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Gay-Related Rejection Sensitivity Scale (GRRS). Scores range from 1 to 36 where higher scores indicate higher stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 13.34 (7.08) | 14.34 (8.38) | 14.48 (7.73)

3. Secondary Outcome: Minority Stress: GRRS
Description: Assessments at 4 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Gay-Related Rejection Sensitivity Scale (GRRS). Scores range from 1 to 36 where higher scores indicate higher stress.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 11.29 (7.05) | 11.33 (7.20) | 11.53 (6.94)

4. Secondary Outcome: Minority Stress: GRRS
Description: Assessments at 8 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Gay-Related Rejection Sensitivity Scale (GRRS). Scores range from 1 to 36 where higher scores indicate higher stress.
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 10.14 (6.14) | 10.51 (7.05) | 11.58 (7.49)

5. Secondary Outcome: Minority Stress: GRRS
Description: Assessments at 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Gay-Related Rejection Sensitivity Scale (GRRS). Scores range from 1 to 36 where higher scores indicate higher stress.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 10.01 (6.79) | 11.07 (7.29) | 10.53 (7.32)

6. Secondary Outcome: Minority Stress: IHS
Description: Assessments at baseline will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Internalized Homonegativity Scale (IHS). The IHS has a range of 1 to 4 with higher scores indicating higher stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 1.90 (0.78) | 1.78 (0.75) | 1.81 (0.70)

7. Secondary Outcome: Minority Stress: IHS
Description: Assessments at baseline, 4, 8, and 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Internalized Homonegativity Scale (IHS). The IHS has a range of 1 to 4 with higher scores indicating higher stress.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 1.73 (0.72) | 1.49 (0.46) | 1.66 (0.62)

8. Secondary Outcome: Minority Stress: IHS
Description: Assessments at 8 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Internalized Homonegativity Scale (IHS). The IHS has a range of 1 to 4 with higher scores indicating higher stress.
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 1.69 (0.67) | 1.44 (0.44) | 1.66 (0.66)

9. Secondary Outcome: Minority Stress: IHS
Description: Assessments at 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Internalized Homonegativity Scale (IHS). The IHS has a range of 1 to 4 with higher scores indicating higher stress.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 1.67 (0.75) | 1.38 (0.42) | 1.53 (0.59)

10. Secondary Outcome: Minority Stress: SOCS
Description: Assessments at baseline will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Sexual Orientation Concealment Scale (SOCS). The SOCS has a range of 1-4 with higher scores indicating higher concealment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 1.84 (0.69) | 1.73 (0.74) | 1.83 (0.76)

11. Secondary Outcome: Minority Stress: SOCS
Description: Assessments at 4 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Sexual Orientation Concealment Scale (SOCS). The SOCS has a range of 1-4 with higher scores indicating higher concealment.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 1.90 (0.70) | 1.79 (0.75) | 1.87 (0.74)

12. Secondary Outcome: Minority Stress: SOCS
Description: Assessments at 8 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Sexual Orientation Concealment Scale (SOCS). The SOCS has a range of 1-4 with higher scores indicating higher concealment.
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 1.94 (0.82) | 1.73 (0.75) | 1.83 (0.76)

13. Secondary Outcome: Minority Stress: SOCS
Description: Assessments at 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Sexual Orientation Concealment Scale (SOCS). The SOCS has a range of 1-4 with higher scores indicating higher concealment.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 1.87 (0.79) | 1.57 (0.73) | 1.83 (0.81)

14. Secondary Outcome: Minority Stress: DERS
Description: Assessments at baseline will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Difficulties of Emotion Regulation Scale (DERS). The DERS has a range of 36 to 172 with higher scores indicating greater difficulty.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 95.39 (20.53) | 98.61 (21.20) | 94.41 (25.20)

15. Secondary Outcome: Minority Stress: DERS
Description: Assessments at 4 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Difficulties of Emotion Regulation Scale (DERS). The DERS has a range of 36 to 172 with higher scores indicating greater difficulty.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 84.84 (21.48) | 94.53 (24.16) | 86.46 (19.62)

16. Secondary Outcome: Minority Stress: DERS
Description: Assessments at 8 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Difficulties of Emotion Regulation Scale (DERS). The DERS has a range of 36 to 172 with higher scores indicating greater difficulty.
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 87.14 (24.29) | 89.34 (21.89) | 86.87 (21.91)

17. Secondary Outcome: Minority Stress: DERS
Description: Assessments at 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Difficulties of Emotion Regulation Scale (DERS). The DERS has a range of 36 to 172 with higher scores indicating greater difficulty.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 85.33 (20.75) | 86.73 (21.21) | 86.09 (20.94)

18. Secondary Outcome: Minority Stress: Brooding
Description: Assessments at baseline will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Brooding Subscale of the Ruminative Response Scale. This scale has a range of 5 to 20 with the higher score indicating greater severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 13.91 (3.08) | 14.25 (3.49) | 13.47 (3.64)

19. Secondary Outcome: Minority Stress: Brooding
Description: Assessments at 4 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Brooding Subscale of the Ruminative Response Scale. This scale has a range of 5 to 20 with the higher score indicating greater severity.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 12.36 (3.21) | 13.20 (3.57) | 13.38 (3.15)

20. Secondary Outcome: Minority Stress: Brooding
Description: Assessments at 8 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Brooding Subscale of the Ruminative Response Scale. This scale has a range of 5 to 20 with the higher score indicating greater severity.
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 12.02 (3.53) | 12.19 (3.45) | 13.14 (3.72)

21. Secondary Outcome: Minority Stress: Brooding
Description: Assessments at 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Brooding Subscale of the Ruminative Response Scale. This scale has a range of 5 to 20 with the higher score indicating greater severity.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 11.55 (3.36) | 12.55 (3.44) | 12.09 (3.50)

22. Secondary Outcome: Minority Stress: Rathus Assertiveness Schedule
Description: Assessments at baseline will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Rathus Assertiveness Schedule. The measure has a range of 39-161 where greater values indicate higher levels of assertiveness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 99.44 (18.77) | 101.39 (20.35) | 99.98 (19.10)

23. Secondary Outcome: Minority Stress: Rathus Assertiveness Schedule
Description: Assessments at 4 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Rathus Assertiveness Schedule. The measure has a range of 39-161 where greater values indicate higher levels of assertiveness.
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 101.87 (15.31) | 105.13 (16.94) | 108.23 (19.62)

24. Secondary Outcome: Minority Stress: Rathus Assertiveness Schedule
Description: Assessments at 8 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Rathus Assertiveness Schedule. The measure has a range of 39-161 where greater values indicate higher levels of assertiveness.
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 104.02 (17.07) | 106.85 (14.94) | 106.47 (18.97)

25. Secondary Outcome: Minority Stress: Rathus Assertiveness Schedule
Description: Assessments at 12 months will be collected to test whether changes in minority stress and mental health precede and statistically mediate the efficacy of ESTEEM. One measurement will come from the Rathus Assertiveness Schedule. The measure has a range of 39-161 where greater values indicate higher levels of assertiveness.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 103.26 (15.32) | 107.47 (15.81) | 108.61 (16.01)

26. Secondary Outcome: Any Condomless Anal Sex Acts
Description: This measure presents the presence (yes/no) of any condomless anal sex (CAS) in the absence of either PrEP or known undetectable viral load of HIV+ primary partners.The Time-Line Follow-Back Interview (TLFB) will be used to assess frequency of HIV risk behavior, including CAS, sex while under the influence of drugs or alcohol, and number of sexual partners, during the previous 3 months.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
Participants
  Yes | 100 | 52 | 101
  No | 0 | 0 | 0
  MISSING | 0 | 0 | 1

27. Secondary Outcome: Any Condomless Anal Sex Acts
Description: as for outcome 26
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 43 | 76
Participants
  Yes | 47 | 24 | 53
  No | 35 | 17 | 21
  MISSING ASSESSMENT | 0 | 2 | 2

28. Secondary Outcome: Any Condomless Anal Sex Acts
Description: as for outcome 26
Time Frame: 12 Months
Population: Participants with completed follow up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
Participants
  Yes | 39 | 26 | 44
  No | 41 | 15 | 36
  MISSING ASSESSMENT | 1 | 1 | 1

29. Secondary Outcome: Safer Sex Self-Efficacy
Description: HIV-relevant information, motivation, and behavioral skills will be assessed using The Safer Sex Self-Efficacy Questionnaire. It is a 13-item measure assessing self-efficacy (confidence) for practicing safer sex. It has demonstrated strong reliability in previous research. Range of scores: 13 - 65. Interpretation: higher scores indicate greater confidence for using condoms during anal sex in the 13 situations listed.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 38.92 (11.73) | 36.69 (12.02) | 38.72 (12.73)

30. Secondary Outcome: Safer Sex Self-Efficacy
Description: as for outcome 29
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 42.83 (12.83) | 37.4 (12.08) | 41.8 (12.69)

31. Secondary Outcome: Safer Sex Self-Efficacy
Description: as for outcome 29
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 42.73 (13.77) | 36.44 (13.11) | 40.32 (10.89)

32. Secondary Outcome: Safer Sex Self-Efficacy
Description: as for outcome 29
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 44.68 (12.32) | 38.55 (13.33) | 41.53 (11.76)

33. Secondary Outcome: Decisional Balance
Description: HIV-relevant information, motivation, and behavioral skills will also be assessed using The Decisional Balance Questionnaire has been used in numerous studies of HIV risk behavior. On this 10-item scale, respondents rate the importance of each of five advantages and disadvantages in their decisions about condom use. Range: 1-5. Interpretation: Scores indicate the importance of each statement upon respondents' decisions to have anal sex with or without condoms. Higher scores on the Pros subscale indicate that pros of having anal sex without a condom (e.g., "sex without a condom is more spontaneous") are rated as important when making the decision to use condoms during anal sex. Higher scores on the Cons subscale indicate that cons of having anal sex without a condom (e.g., "I could get infected with HIV if I have sex without a condom") are rate as important when making the decision to use condoms during anal sex.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale
  Pros Subscale | 2.62 (0.81) | 2.8 (0.74) | 2.66 (0.77)
  Cons Subscale | 3.26 (0.81) | 3.16 (0.81) | 3.24 (0.8)

34. Secondary Outcome: Decisional Balance
Description: as for outcome 33
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale
  Pros Subscale | 2.45 (0.83) | 2.71 (0.7) | 2.65 (0.85)
  Cons Subscale | 3.17 (0.85) | 3.19 (0.83) | 3.19 (0.84)

35. Secondary Outcome: Decisional Balance
Description: as for outcome 33
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale
  Pros Subscale | 2.31 (0.83) | 2.83 (0.65) | 2.44 (0.68)
  Cons Subscale | 3.12 (0.9) | 3.08 (0.82) | 3.02 (0.84)

36. Secondary Outcome: Decisional Balance
Description: as for outcome 33
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale
  Pros Subscale | 2.46 (0.88) | 2.71 (0.77) | 2.46 (0.68)
  Cons Subscale | 3.17 (0.9) | 3.26 (0.83) | 3.0 (0.85)

37. Secondary Outcome: Depression: HAM-D
Description: To determine depression symptom severity, interviewers will complete the Hamilton Rating Scale for Depression (HAM-D). The HAM-D has a range of 0-32 where higher scores indicate greater levels of depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 16.13 (6.26) | 15.87 (6.75) | 15.25 (6.83)

38. Secondary Outcome: Depression: HAM-D
Description: as for outcome 37
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 10.20 (6.13) | 9.93 (6.82) | 10.51 (7.02)

39. Secondary Outcome: Depression: HAM-D
Description: as for outcome 37
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 9.81 (6.04) | 9.57 (6.20) | 11.72 (6.39)

40. Secondary Outcome: Depression: HAM-D
Description: as for outcome 37
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 9.95 (6.34) | 11.49 (8.86) | 10.73 (6.68)

41. Secondary Outcome: Depression: BSI GSI
Description: The Global Severity Index (GSI) of the 18-item Brief Symptom Inventory (BSI) provides a mean score across depression, anxiety, and somatization subscales, and assesses psychological distress (e.g., "feeling nervousness or shakiness inside") on a 5-point scale from 0 (not at all) to 4 (extremely).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
score on a scale | 1.23 (0.62) | 1.29 (0.62) | 1.31 (0.67)

42. Secondary Outcome: Depression: BSI GSI
Description: as for outcome 41
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
score on a scale | 0.66 (0.60) | 0.86 (0.73) | 0.77 (0.66)

43. Secondary Outcome: Depression: BSI GSI
Description: as for outcome 41
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
score on a scale | 0.60 (0.54) | 0.69 (0.61) | 0.80 (0.60)

44. Secondary Outcome: Depression: BSI GSI
Description: as for outcome 41
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
score on a scale | 0.65 (0.63) | 0.70 (0.69) | 0.76 (0.64)

45. Secondary Outcome: Substance Use: SIP-AD
Description: Short Inventory of Problems - Alcohol and Drugs (SIP-AD; Allensworth-Davies et al., 2012; Blanchard et al., 2003). SIP-AD is a 15-item scale in which the sum of "yes" responses indicates participants' past-3-month consequences of alcohol and drug use (e.g., "I have failed to do what is expected of me because of my drinking/drug use"). Higher scores indicate greater substance use with a range of 0-15.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
units on a scale | 4.95 (4.42) | 4.71 (4.06) | 4.52 (4.41)

46. Secondary Outcome: Substance Use: SIP-AD
Description: as for outcome 45
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 83 | 43 | 76
units on a scale | 3.21 (4.19) | 4.29 (3.98) | 3.34 (3.94)

47. Secondary Outcome: Substance Use: SIP-AD
Description: as for outcome 45
Time Frame: 8 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 36 | 77
units on a scale | 2.72 (3.33) | 3.75 (4.17) | 3.38 (4.07)

48. Secondary Outcome: Substance Use: SIP-AD
Description: as for outcome 45
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 81 | 42 | 81
units on a scale | 2.51 (3.54) | 3.83 (4.18) | 2.79 (3.61)

49. Secondary Outcome: Any Pre-Exposure Prophylaxis (PrEP) Use
Description: Participants will be asked if they had used PrEP in the last 3 months.
Time Frame: Baseline
Population: Participants that either completed or partially completed the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 101
Participants
  No, I have never taken HIV PrEP | 82 | 41 | 87
  Yes, I am currently taking HIV PrEP | 0 | 0 | 1
  I am not currently taking HIV PrEP, but I have taken PrEP within the past 3 months | 3 | 3 | 3
  I am not currently taking HIV PrEP, but I have taken PrEP more than 3 months ago | 15 | 8 | 10

50. Secondary Outcome: Any Pre-Exposure Prophylaxis (PrEP) Use
Description: Participants will be asked if they had used PrEP in the last 3 months.
Time Frame: 4 Months
Population: Participants that either completed or partially completed the interview, MISSING used for those that either dropped our or partially completed the interview.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 82 | 43 | 76
Participants
  No, I have never taken HIV PrEP | 63 | 25 | 54
  Yes, I am currently taking HIV PrEP | 10 | 13 | 10
  I am not currently taking HIV PrEP, but I have taken PrEP within the past 3 months | 2 | 0 | 1
  I am not currently taking HIV PrEP, but I have taken PrEP more than 3 months ago | 7 | 4 | 9
  MISSING ASSESSMENT | 0 | 1 | 2

51. Secondary Outcome: Any Pre-Exposure Prophylaxis (PrEP) Use
Description: Participants will be asked if they had used PrEP in the last 3 months.
Time Frame: 8 Months
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 101
Participants
  No, I have never taken HIV PrEP | 56 | 21 | 44
  Yes, I am currently taking HIV PrEP | 11 | 9 | 20
  I am not currently taking HIV PrEP, but I have taken PrEP within the past 3 months | 7 | 2 | 2
  I am not currently taking HIV PrEP, but I have taken PrEP more than 3 months ago | 8 | 4 | 11
  MISSING | 18 | 16 | 25

52. Secondary Outcome: Any Pre-Exposure Prophylaxis (PrEP) Use
Description: Participants will be asked if they had used PrEP in the last 3 months.
Time Frame: 12 Months
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 101
Participants
  No, I have never taken HIV PrEP | 50 | 22 | 44
  Yes, I am currently taking HIV PrEP | 11 | 7 | 20
  I am not currently taking HIV PrEP, but I have taken PrEP within the past 3 months | 7 | 5 | 3
  I am not currently taking HIV PrEP, but I have taken PrEP more than 3 months ago | 13 | 8 | 14
  MISSING | 19 | 10 | 21

53. Other Pre Specified Outcome: HIV Test
Description: Orasure Rapid HIV-1/2 Antibody Test will be used to test participants for HIV at Baseline.
Time Frame: Baseline
Population: Participants with complete and valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
Participants
  Negative | 100 | 52 | 102
  Preliminary Positive | 0 | 0 | 0

54. Other Pre Specified Outcome: HIV Test
Description: Orasure Rapid HIV-1/2 Antibody Test will be used to test participants for HIV at 12 months.
Time Frame: 12 Months
Population: Participants with complete and valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 76 | 39 | 76
Participants
  Negative | 73 | 39 | 75
  Preliminary Positive | 3 | 0 | 1

55. Other Pre Specified Outcome: Gonorrhea Test
Description: Oral, rectal and urine samples will be collected to test participants for Gonorrhea at Baseline.
Time Frame: Baseline
Population: Participants with complete and valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
Participants
  Throat: Non-reactive | 94 | 48 | 97
  Throat: Reactive | 5 | 4 | 4
  Throat: Inconclusive | 0 | 0 | 1
  Throat: Not Assessed | 1 | 0 | 0
  Rectal: Non-reactive | 95 | 49 | 99
  Rectal: Reactive | 5 | 3 | 1
  Rectal: Inconclusive | 0 | 0 | 1
  Rectal: Not Assessed | 0 | 0 | 1
  Urine: Non-reactive | 100 | 52 | 102
  Urine: Reactive | 0 | 0 | 0
  Urine: Inconclusive | 0 | 0 | 0
  Urine: Not Assessed | 0 | 0 | 0

56. Other Pre Specified Outcome: Gonorrhea Test
Description: Oral, rectal and urine samples will be collected to test participants for Gonorrhea at 12 months.
Time Frame: 12 Months
Population: Participants with complete and valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 74 | 38 | 75
Participants
  Throat: Non-reactive | 71 | 36 | 73
  Throat: Reactive | 2 | 2 | 2
  Throat: Inconclusive | 0 | 0 | 0
  Throat: Not assessed | 1 | 0 | 0
  Rectal: Non-reactive | 67 | 35 | 73
  Rectal: Reactive | 5 | 3 | 2
  Rectal: Inconclusive | 0 | 0 | 0
  Rectal: Not assessed | 2 | 0 | 0
  Urine: Non-reactive | 74 | 38 | 75
  Urine: Reactive | 0 | 0 | 0
  Urine: Inconclusive | 0 | 0 | 0
  Urine: Not assessed | 0 | 0 | 0

57. Other Pre Specified Outcome: Chlamydia Test
Description: Oral, rectal and urine samples will be collected to test participants for Chlamydia at Baseline.
Time Frame: Baseline
Population: Participants with complete and valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 100 | 52 | 102
Participants
  Throat: Non-reactive | 97 | 50 | 96
  Throat: Reactive | 2 | 2 | 5
  Throat: Inconclusive | 0 | 0 | 1
  Throat: Not assessed | 1 | 0 | 0
  Rectal: Non-reactive | 97 | 48 | 90
  Rectal: Reactive | 3 | 4 | 10
  Rectal: Inconclusive | 0 | 0 | 1
  Rectal: Not assessed | 0 | 0 | 1
  Urine: Non-reactive | 99 | 51 | 101
  Urine: Reactive | 1 | 1 | 1
  Urine: Inconclusive | 0 | 0 | 0
  Urine: Not assessed | 0 | 0 | 0

58. Other Pre Specified Outcome: Chlamydia Test
Description: Oral, rectal and urine samples will be collected to test participants for Chlamydia at 12 months.
Time Frame: 12 Months
Population: Participants with complete and valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
Number analyzed (Participants) | 74 | 38 | 75
Participants
  Throat: Non-reactive | 72 | 38 | 75
  Throat: Reactive | 1 | 0 | 0
  Throat: Inconclusive | 0 | 0 | 0
  Throat: Not assessed | 1 | 0 | 0
  Rectal: Non-reactive | 69 | 34 | 74
  Rectal: Reactive | 3 | 4 | 1
  Rectal: Inconclusive | 0 | 0 | 0
  Rectal: Not assessed | 2 | 0 | 0
  Urine: Non-reactive | 74 | 38 | 75
  Urine: Reactive | 0 | 0 | 0
  Urine: Inconclusive | 0 | 0 | 0
  Urine: Not assessed | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Severe Adverse Events were assessed systematically using the Brief Symptom inventory (BSI) and Suicidal Ideation Attributes Scale (SIDAS) during in-office assessments at 4MFU, 8MFU and 12MFU. Active suicidality also assessed through participant self-disclosure during therapy or during semi-structured clinical interviews (HAMD) during follow-up visits.
Arm/Group | ESTEEM | Voluntary Counselling and Testing (VCT) | Community Mental Health Treatment (CMHT)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/52 | 0/102
Serious Adverse Events (participants affected / at risk) | 4/100 | 0/52 | 1/102
Other Adverse Events (participants affected / at risk) | 0/100 | 0/52 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESTEEM (N=100) | Voluntary Counselling and Testing (VCT) (N=52) | Community Mental Health Treatment (CMHT) (N=102)
Active Suicidality (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT02929069/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT02929069/SAP_001.pdf